CLINICAL TRIAL: NCT00693901
Title: Parks and Physical Activity in Diverse Communities
Brief Title: Influence of Public Parks on Physical Activity Levels of Diverse Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 499; R01HL083869 (NIH)
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Community-Based Participatory Research

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Parks will be assigned to the community-based participatory research condition.
  Interventions: Behavioral: Community-based participatory research (CBPR)
- 2 (Active Comparator): Parks will be assigned to the director-only condition.
  Interventions: Behavioral: Director-only
- 3 (No Intervention): Parks will be assigned to the control condition and will receive no intervention.

INTERVENTIONS:
Behavioral: Community-based participatory research (CBPR) — CBPR will involve park advisory boards and community members in the research process, including the park assessments and data analysis. The assessment research will be used to inform use of discretionary funds for park programming and facilities in the hopes of increasing community physical activity. Park directors will be provided with analysis of descriptive information and community feedback to help improve outreach, park programming, and features to attract more park users and increase physical activity.
  Arms: 1
Behavioral: Director-only — Park directors will be provided with descriptive information on park use and community feedback. They will also receive assistance on how to improve outreach, programming, and park features that will increase park use and physical activity. These parks will not take part in any assessments.
  Arms: 2

SUMMARY:
Engaging in physical activity is an important health behavior for maintaining good health and preventing disease. Public parks offer community members readily accessible areas for recreation and exercise. Modifying park programs and facilities to meet the specific needs of community members may encourage people to engage in more physical activity. Furthermore, using feedback from the community might be the best way to determine how park funds should be allocated for modifications. This study will compare two approaches to park programming and will determine which approach is best at increasing physical activity within the community.

DETAILED DESCRIPTION:
Regular physical activity, such as walking, running, or biking, is known to have substantial health benefits. Exercise is important not only in weight management, but also in reducing the risk of certain diseases and promoting psychological well being. In fact, each year about 1.9 million deaths are attributed to physical inactivity, making programs to promote increased physical activity a public health priority. Public parks are easily accessible recreational areas, and they provide beneficial places to implement programs that encourage physical activity among community members. Using information on park use and assessments of community feedback may help improve park outreach, programming, and features aimed to increase physical activity in the community. This study will compare two approaches to park programming and will determine which approach is best at increasing physical activity within the community. The first approach is CBPR, a research program that involves community members in scientific and systematic park assessments that are then analyzed to guide park programming. The second approach simply provides park utilization and community feedback data to park directors to guide park programming.

Park participation in this study will last 1 year. Participating parks will be assigned randomly to one of three conditions:

* Parks assigned to Condition 1 will participate in CBPR, which will include assessments of observations and surveys about park programs and facilities. Anonymous members of the surrounding community will be involved in the assessments, which will be conducted at baseline and Year 1.
* Parks assigned to Condition 2 will receive the director-only condition. These parks will not take part in any assessments, but park directors will be provided with park utilization data, community feedback, and ways to improve park features to increase physical activity.
* Parks assigned to Condition 3 will receive the control condition and will not take part in the assessments or be provided with park utilization data and community feedback.

Administrative data about parks and park functions will also be collected from all participating parks.

ELIGIBILITY:
Inclusion Criteria:

* Neighborhood park with an advisory board
* Park director who is willing to participate

Exclusion Criteria:

* Park that is NOT a neighborhood park

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Composite measure of energy expenditure at public parks | Measured at Year 5

SECONDARY OUTCOMES:
Number of park users | Measured at Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Cohen, MD, MPH, Principal Investigator — RAND
Locations (1):
- RAND, Santa Monica, California, United States